CLINICAL TRIAL: NCT00160069
Title: Phase II Study to Investigate the Efficacy and Safety of ZK 219477 as Second Line Therapy in Patients With Stage IIIB or Stage IV Non Small Cell Lung Cancer (NSCLC)
Brief Title: Safety and Efficacy Study of a New Chemotherapy Agent to Treat Non-small-cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 91374; 2005-000586-19 (EudraCT Number); 307971 (Other: Company Internal ID)
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Carcinoma, Non Small Cell Lung
Keywords: Stage IIIB or stage IV non-small-cell lung cancer.
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — sagopilone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Drug: Sagopilone (BAY86-5302, ZK 219477)
- Arm 2 (Experimental)
  Interventions: Drug: Sagopilone (BAY86-5302, ZK 219477)
- Arm 3 (Experimental)
  Interventions: Drug: Sagopilone (BAY86-5302, ZK 219477)

INTERVENTIONS:
Drug: Sagopilone (BAY86-5302, ZK 219477) — 16 mg/m2, 3-hour infusion, every 3 weeks
  Arms: Arm 1
Drug: Sagopilone (BAY86-5302, ZK 219477) — 22 mg/m2, 30-min infusion, every 3 weeks
  Arms: Arm 2
Drug: Sagopilone (BAY86-5302, ZK 219477) — 22 mg/m2, 3-hour infusion, every 3 weeks
  Arms: Arm 3

SUMMARY:
Phase 2 study to investigate the efficacy and tolerability of epothilone ZK 219477 in patients with stage IIIb or stage IV non-small-cell lung cancer.

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer Schering Pharma AG, Germany.Bayer Schering Pharma AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Non-small-cell lung cancer
* Only one previous chemotherapy with a platinum-containing drug
* Use of highly effective birth control methods in females of child-bearing potential

Exclusion Criteria:

* No more than 1 previous chemotherapy for advanced disease
* Previous participation in another trial within the last 4 weeks
* Breast feeding
* Active infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2005-08; Primary Completion 2008-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variable is defined as Proportion of patients with either CR or PR as 'best overall response'. Tumor assessment is performed according to RECIST criteria. | Tumor evaluation (MRI or scan) every 2 cycles until disease progression.

SECONDARY OUTCOMES:
Secondary objectives : investigate the safety and tolerability of ZK 219477 | Continuously

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (15):
- Germany (15):
  - Löwenstein, Baden-Wurttemberg
  - Augsburg, Bavaria
  - Gauting, Bavaria
  - Nuremberg, Bavaria
  - Hamburg, Hamburg
  - Frankfurt am Main, Hesse
  - Greifswald, Mecklenburg-Vorpommern
  - Stralsund, Mecklenburg-Vorpommern
  - Leipzig, Saxony
  - Halle, Saxony-Anhalt
  - Magdeburg, Saxony-Anhalt
  - Großhansdorf, Schleswig-Holstein
  - Berlin, State of Berlin
  - Bremen
  - Ebensfeld

REFERENCES:
- [Result] Heigener DF, von Pawel J, Eschbach C, Brune A, Schmittel A, Schmelter T, Reck M, Fischer JR. Prospective, multicenter, randomized, independent-group, open-label phase II study to investigate the efficacy and safety of three regimens with two doses of sagopilone as second-line therapy in patients with stage IIIB or IV non-small-cell lung cancer. Lung Cancer. 2013 Jun;80(3):319-25. doi: 10.1016/j.lungcan.2013.02.007. Epub 2013 Mar 20. PMID 23522488
- See also: Click here and search for Bayer product information provided by the EMA — http://www.clinicaltrialsregister.eu